CLINICAL TRIAL: NCT01969409
Title: Autoantibody Reduction Therapy in Patients With Idiopathic Pulmonary Fibrosis (ART-IPF)
Brief Title: Autoantibody Reduction Therapy in Patients With Idiopathic Pulmonary Fibrosis
Acronym: ART-IPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Steven R. Duncan, MD, Priniciple Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL119960
Record Dates: First submitted 2013-10-17; First posted 2013-10-25 (Estimated); Results first posted 2021-11-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Ambulatory IPF
Keywords: Lung; Fibrosis
MeSH Terms: conditions — Fibrosis | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): These subjects will receive i.v. placebo (5% dextrose in water) administered identically to the rituximab.
  Interventions: Drug: Placebo
- Rituximab (Experimental): Rituximab i.v. given on two occasions, with 14 days between doses.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — i.v. rituximab given on two occasions 14 days apart.
  Arms: Rituximab
Drug: Placebo — Subjects randomized to placebo will receive two i.v. doses of 5% dextrose in water (D5W) in the same schedule as the rituximab subjects. The D5W and rituximab preparations will be indistinguishable.
  Other Names: Placebo (D5W) i.v.
  Arms: Placebo

SUMMARY:
Recent research studies have suggested that proteins called antibodies that are produced by the immune system might be involved in the lung damage of idiopathic pulmonary fibrosis (IPF). Antibodies produced by the immune system normal help to fight infections by attacking bacteria and viruses without harming our own tissues. In patients with IPF, there is evidence that certain antibodies (called autoantibodies) attack the lung and contributes to the injury and scarring that occurs in IPF. Our recent studies have found that many IPF patients appear to have excessive autoantibody levels in blood and lungs that might make their disease worse.

Rituximab is a medication approved by the Food and Drug Administration (FDA) for the treatment of autoantibody diseases such as rheumatoid arthritis. Rituximab works by destroying B cells, a type of white blood cell, called a B-lymphocyte, which produce autoantibodies. In this research study, rituximab will be given into a vein to reduce the autoantibody levels that we believe might be contributing to the lung damage in IPF.

This study is being conducted to determine if rituximab provides beneficial effects for IPF patients by decreasing further lung injury.

DETAILED DESCRIPTION:
This is a double-blinded, Phase II trial in which 58 ambulatory IPF patients at any of four medical centers (University of Pittsburgh, University of Chicago, Geisinger Medical Center, and Temple University) will be randomized equally to 1. placebo or 2. two doses of rituximab 1 gm i.v., with a 14 day interval inbetween doses.

Subjects will be followed for 9 months.

ELIGIBILITY:
Inclusion Criteria:

Ambulatory patients with a diagnosis of IPF, not established >5 years from the enrollment date, that fulfills American Thoracic Society (ATS)/European Thoracic Society (ETS) Consensus Criteria.

Ability and willingness to give informed consent. Presence of autoantibodies against Hepatoma-2 (HEp-2) cells, the assay for the primary endpoint.

Age 50-85 y.o.

Exclusion Criteria:

Diagnoses of current infection, proven or suspected by participating physicians based upon their clinical assessments.

Presence of active hepatitis B or C, or HIV infection. Presence of positive CONVENTIONAL autoimmune serologic tests, e.g., Antinuclear Antibodies (ANA), Rheumatoid Factor (RF), Anti-Ro, Anti-LA, Anti-Ribonucleoprotein Antibodies (RNP), Anti-Jo-1.

History of reaction to murine-derived products or any of the trial medications, or prior exposures to human-murine chimeric antibodies.

Malignancy, excluding basal or squamous cell skin cancer and low-risk prostate cancer, defined as stage T1 or T2a with Prostate-Specific Antigen (PSA) less than 10 ng/dl.

Unwillingness to complete post-treatment surveillance for 9 months. Diagnosis of major morbidities (aside from IPF) expected to interfere with subjects' study participation for 9 months.

Treatment for >5 days within the preceding month with >10 mg. prednisone (or equivalent corticosteroid) or any treatment during the preceding month with a potent cellular immunosuppressant (e.g., cyclophosphamide, methotrexate, mycophenolate, azathioprine, calcineurin inhibitors, etc.).

Uncontrolled diabetes or hypertension that preclude safe treatment with methylprednisolone.

Concurrent participation in other experimental trials.

Pregnancy or unwillingness to use contraception during the duration of the study among female participants with child-bearing potential.

Ratio of forced expiratory volume in 1 second to forced vital capacity (FEV1/FVC) <70% of predicted values.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Duncan, MD, Principal Investigator — University of Alabama at Birmingham
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnestoa, Minneapolis, Minnesota
  - Geisinger Medical Center, Danville, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Rituximab
Started | 28 | 30
Completed | 25 | 26
Not Completed | 3 | 4
Not completed — Death | 2 | 2
Not completed — Transplant | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rituximab | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (7) | 68 (7) | 69 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 23 | 23 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 30 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 58

OUTCOME MEASURES:

1. Primary Outcome: Autoantibodies to Human Epidermoid (HEp)-2 Cells
Description: Titers of anti-HEp-2 autoantibodies, by indirect immunofluorescence assays (IFA) over 9 months, month 9 reported. Titers represent the highest dilution of patient plasma wherein the autoantibodies can be detected. Higher titers denote greater autoantibody concentrations.
Time Frame: baseline to 9 months
Population: 7 not analyzed: 4 deaths, 2 transplants, 1 dropout
Measure: Mean (Standard Error); unit: titer
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 25 | 26
titer | 288 (63) | 177 (29)

2. Secondary Outcome: Changes in Anti-Heat Shock Protein 70 (HSP70) Autoantibodies
Description: Changes of anti-HSP70 plasma concentrations as determined by ELISA, month 9 reported. The result is expressed as optical density (OD) units. The greater the number; the more autoantibody.
Time Frame: baseline to 9 months
Population: 7 not analyzed: 4 deaths, 2 transplants, 1 dropout
Measure: Mean (Standard Error); unit: OD units
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 25 | 26
OD units | 1.0 (0.13) | 0.83 (0.08)

3. Secondary Outcome: Changes in Forced Vital Capacity (FVC)
Description: FVC values over the observation period will be measured by spirometry, month 9 reported.
Time Frame: baseline thru 9 months
Population: 7 not analyzed: 4 deaths, 2 transplants, 1 dropout
Measure: Mean (Standard Error); unit: liters
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 25 | 26
liters | 2.6 (0.14) | 2.5 (0.16)

4. Secondary Outcome: Number of Adverse Events (AE)
Description: AE in the two treatment arms will be compared. Serious adverse events, as defined by national toxicity scale.
Time Frame: during the 9 months of observation
Population: Data not complete in 7 due to 4 deaths, 2 transplants, 1 dropout
Measure: Number; unit: serious adverse events
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 25 | 26
serious adverse events | 7 | 12

5. Secondary Outcome: Number of Acute Exacerbations
Description: The number of acute exacerbations, defined using consensus criteria (new/worsened hypoxemia and dyspnea, with characteristic radiographic changes within the last 30 days).
Time Frame: during the study duration of 9 months
Population: Data from 7 incomplete: 4 deaths, 2 transplants, 1 dropout
Measure: Number; unit: acute exacerbations
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 25 | 26
acute exacerbations | 1 | 2

6. Secondary Outcome: Absolute Survival Percentage
Description: Absolute survival in the two arms calculated by actuarial methods (Kaplan-Meier). These result in percent survival denoted as means and +/- standard error (these are detailed in the outcome table below).
Time Frame: during 9 months of observation
Population: 1 dropout (censored event)
Measure: Mean (Standard Error); unit: percent of participants
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 28 | 30
percent of participants | 93 (5) | 93 (5)

7. Secondary Outcome: Transplant-Free Survival
Description: Actuarial transplant-free survival in the two arms, calculated by actuarial methods (Kaplan-Meier).
  These result in percent survival denoted as means and +/- standard error (these are detailed in the outcome table below).
Time Frame: during 9 months of observation
Population: 1 dropout
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 28 | 29
percentage of participants | 89 (6) | 90 (6)

8. Secondary Outcome: Hospitalizations
Description: The number of hospitalizations in the two arms will be compared.
Time Frame: during 9 months of observation
Population: incomplete data on 1 dropout
Measure: Number; unit: number of admissions
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 28 | 30
number of admissions | 6 | 12

ADVERSE EVENTS:
Time Frame: Baseline to 9 months
Arm/Group | Placebo | Rituximab
All-Cause Mortality (participants affected / at risk) | 2/28 | 2/30
Serious Adverse Events (participants affected / at risk) | 5/28 | 9/30
Other Adverse Events (participants affected / at risk) | 21/28 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Rituximab (N=30)
Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Pneumonia
Infection (Gastrointestinal disorders) | 0 (0) | 2 (2) — Appendicitis Colitis
Worsening respiratory function (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) — Increased dyspnea without acute exacerbation
cerebral vascular accident (Nervous system disorders) | 1 (1) | 0 (0) — stroke
syncope (Nervous system disorders) | 1 (1) | 0 (0) — syncope
Acute exacerbation of idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — Acute exacerbation
Myocardial Infarct (Cardiac disorders) | 0 (0) | 2 (2) — myocardial infarct
Right ventricular failure (Cardiac disorders) | 2 (2) | 0 (0) — Right heart failure
carotid revascularization (Nervous system disorders) | 0 (0) | 1 (1) — carotid artery stint
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Rituximab (N=30)
flushing (General disorders) | 2 (2) | 2 (3) — flushing
fever (General disorders) | 1 (1) | 2 (3) — fever self reported
dry mouth (General disorders) | 4 (7) | 3 (6) — dry mouth
Infection unspecified (mild) (Infections and infestations) | 2 (2) | 0 (0) — infection
chest tightness (Cardiac disorders) | 2 (2) | 0 (0) — chest tightness, Not Otherwise Specified (NOS)
arrhythmia (Cardiac disorders) | 3 (3) | 0 (0) — mild, NOS
Hypertension (Cardiac disorders) | 2 (3) | 2 (5) — blood pressure elevated greater than usual
palpitations (Cardiac disorders) | 0 (0) | 2 (2) — self reported palpitations NOS
Pruritis (Skin and subcutaneous tissue disorders) | 2 (5) | 3 (3) — pruritis
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 7 (7) — skin rash NOS
Brusing (Surgical and medical procedures) | 2 (2) | 1 (1) — Ecchymosis
abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3) — abdominal pain self limited and NOS
Anorexia (Gastrointestinal disorders) | 2 (3) | 3 (3) — loss of appetite
Diarrhea (Gastrointestinal disorders) | 4 (7) | 5 (5) — diarrhea
Nausea (Gastrointestinal disorders) | 4 (5) | 6 (7) — nausea with or without vomiting
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) — elevated blood sugar greater than baseline
Anxiety (Nervous system disorders) | 2 (3) | 0 (0) — anxiety
Dizzyness (Nervous system disorders) | 3 (8) | 2 (3) — dizziness self reported
Fatigue (Nervous system disorders) | 4 (7) | 3 (6) — self reported fatigue NOS
Headache (Nervous system disorders) | 3 (4) | 5 (9) — headache
Insomnia (Nervous system disorders) | 4 (5) | 5 (5) — trouble sleeping
cough (Respiratory, thoracic and mediastinal disorders) | 7 (15) | 10 (12) — Cough greater than baseline
Post-nasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) — post-nasal discharge
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (18) | 5 (18) — Shortness of breath greater than baseline not attributable to acute exacerbations, pneumonia, or causes other than idiopathic pulmonary fibrosis
dry eyes (Eye disorders) | 2 (3) | 0 (0) — dry eyes, self-limited
Backache (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) — back pain, self limited
Muscle pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) — Muscle pain other than backache (self limited)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — self limited joint stiffness
urinary tract infection (Renal and urinary disorders) | 1 (1) | 2 (4) — urinary tract infection documented by culture or suspected
Tooth infection (Infections and infestations) | 0 (0) | 2 (2) — tooth infection self-reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT01969409/Prot_SAP_000.pdf